CLINICAL TRIAL: NCT00502879
Title: A Randomized, Open-Label, Single-Dose Administration, Parallel-Group Study of the Pharmacokinetics of Etanercept, 25mg or 50 mg, Administered Subcutaneously to Healthy Chinese Male Subjects
Brief Title: Study Evaluating Etanercept 25mg or 50mg Administered Subcutaneously to Healthy Chinese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0881A1-1109
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Last update posted 2007-12-06 (Estimated); Status verified 2007-12

CONDITIONS: Healthy
MeSH Terms: interventions — Etanercept

INTERVENTIONS:
Drug: Enbrel (etanercept)

SUMMARY:
The primary purpose of this study is to assess the pharmacokinetics of etanercept in healthy Chinese male subjects. Safety and tolerability data will also be obtained.

ELIGIBILITY:
1. Men, aged 18 to 45 years, of Chinese descent and living in China.
2. Body mass index in the range of 18.0 to 30.0 kg/meter squared and body weight equal to or greater than 50 kg.
3. Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, chest x-ray, and 12-lead electrocardiogram (ECG).
4. Have a high probability for compliance with and completion of the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2007-07; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
To assess the pharmacokinetics of etanercept in healthy Chinese male subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For China: medinfo@wyeth.com
Locations (1):
- Beijing, China